CLINICAL TRIAL: NCT01595750
Title: Randomized, Double-blind, Placebo-controlled Study to Evaluate the Effect of Roflumilast on Endothelial Function in Patients With Chronic Obstructive Pulmonary Disease
Acronym: REVASC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Spanish Research Center for Respiratory Diseases (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIB-ROF-2011-01; 2011-005047-27 (EudraCT Number)
Record Dates: First submitted 2012-05-09; First posted 2012-05-10 (Estimated); Last update posted 2012-05-10 (Estimated); Status verified 2012-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Post-bronchodilator FEV1<70% reference; Chronic bronchitis; Presence of estavlished CVD,; CVD equivalent or diabetes mellitus
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Roflumilast (Active Comparator): Roflumilast 500 mcg
  Interventions: Drug: Roflumilast 500

INTERVENTIONS:
Drug: Roflumilast 500 — Roflumilast 500 mcg , 12 weeks of treatment
  Arms: Roflumilast
Drug: Placebo — Placebo 500 mcg , 12 weeks of treatment
  Arms: Placebo

SUMMARY:
REVASC is a randomized, double-blind, placebo-controlled study which will involve 150 patients with chronic bronchitis and COPD diagnosed cardiovascular disease. The recruitment period beginimg in the coming weeks, will last nine months. Patients included in the study will receive treatment for three months with roflumilast 500 mg (75 patients) or placebo (75 patients) in a randomized manner. The CIBERES, as promoter of this study is expected to release final results for the third quarter of 2013.

Eight centers in Madrid will be involved in this clinical trial: Fundación Jiménez Díaz, Hospital La Princesa, Hospital Gregorio Maranon Hospital Clinico San Carlos, Hospital La Paz, Hospital Ramón y Cajal Hospital Doce de Octubre and Hospital Puerta del Hierro.

Roflumilast is a potent phosphodiesterase-4 inhibitor (PDE4). Its clinical efficacy has been studied in an extensive clinical program involving over 12,000 patients with COPD. In these studies, roflumilast (in combination with long-acting bronchodilators) reduced the number of exacerbations and improved lung function, especially in those patients with associated chronic bronchitis.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* 55-75 years of age
* Current and former smokers >20 cigarettes pack-yr (if former smokers withdrawn >1 year)
* Diagnosis COPD (GOLD criteria1 for more than a year before V0)
* Presence of chronic bronchitis (cough and/or expectoration for more that 3 months/yr for more than 2 consecutive yrs. in the absence of other potential cause)
* Post-bronchodilator FEV1<70% reference
* Presence of established CVD, CVD equivalent or diabetes mellitus
* Presence of chronic systemic inflammation, determined on:

  1. Serum CRP ≥ 2 and < 10 mg/l or
  2. Serum fibrinogen > 518 mg/dl and Leucocytes > 8,6*106 /mm3

Exclusion Criteria:

* Episode of COPD exacerbation and/or COPD treatment change during the last 2 months before V0
* History of asthma, significant residual lung lesions or bronchiectasis on chest x-ray
* Apnea-hypopnea syndrome
* Poorly controlled CVD risk factors (Table 2) and/or change in their treatment during the last 3 months before V0
* Clinically significant cardiac arrhythmias or valve disease
* Severe concomitant immunological, inflammatory, infectious or neoplastic diseases
* Moderate or severe hepatic insufficiency (B or C class, following Child-Pugh scale)
* Severe neurologic and/or psychiatric disorder, including depression with suicidal ideas
* Alcohol and/or drug abuse during the last 12 months before V0
* Hypersensitivity to roflumilast or to any of its excipients
* Pregnancy or potential pregnancy
* Participation in other clinical trial during the last 30 days before V0
* Language difficulties to follow the instructions of the study

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2012-05; Primary Completion 2012-07 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Endotelial function | 12 weeks

SECONDARY OUTCOMES:
Arterial siffness | 12 weeks
Serum and plasma inflammation markers: (CRP, fibrinogen, leucocytes, interleukin (IL)-8, IL-6, IL-10, tumor necrosis factor alpha (TNFα), sICAM-1, MCP-1, PARC/CCL-18) | 12 weeks
Serum oxidatrive stress markers: MPO, TRX | 12 weeks
Serum endothelial dysfunction markers:TWEAKs, FasL, ADMA | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Julio Ancochea, Principal Investigator — Hospital Universitario La Princesa; Carlos Álvarez, Principal Investigator — Hospital Universitario Doce de Octubre; Pilar De Lucas, Principal Investigator — Hospital General Universitario Gregorio Marañón; Myriam Calle, Principal Investigator — Hospital Clínico Universitario San Carlos; Salvador Díaz, Principal Investigator — Hospital Universitario Ramón y Cajal; Francisco García, Principal Investigator — Hospital Universitario La Paz; Rosa Malo, Principal Investigator — Hospital Universitario Puerta de Hierro; Germán Peces-Barba, Principal Investigator — Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz
Locations (1):
- Spanish Research Center for Respiratory Diseases, Bunyola, Balearic Island, Spain